CLINICAL TRIAL: NCT04324463
Title: Anti-Coronavirus Therapies to Prevent Progression of COVID-19, a Randomized Trial
Brief Title: Anti-Coronavirus Therapies to Prevent Progression of Coronavirus Disease 2019 (COVID-19) Trial
Acronym: ACTCOVID19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRI.ACT.COVID19
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Coronavirus; Severe Acute Respiratory Syndrome
Keywords: COVID-19; coronavirus; interferon; colchicine; aspirin; rivaroxaban; anti-inflammatory; antithrombotic; anti-viral
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; COVID-19 | interventions — Colchicine; Interferon-beta; Aspirin; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Open-label, parallel group, factorial, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Colchicine (Experimental): Outpatients:
  0.6 mg twice daily for 3 days, then 0.6 mg once daily for 25 days (total 28 days).
  Inpatients:
  1.2 mg followed by 0.6 mg 2 hours later, then 0.6 mg twice daily for 28 days.
  (*Depending on availability, 0.6 mg tablets can be substituted by 0.5 mg tablets for a regimen in outpatients of 0.5 mg twice daily for 3 days, then 0.5 mg once daily for 25 days [total 28 days]; and in inpatients of 1.0 mg followed by 0.5 mg 2 hours later, then 0.5 mg twice daily for 28 days).
  Interventions: Drug: Colchicine
- Interferon Beta [This arm is now closed to recruitment] (Experimental): Inpatients Only:
  0.25 mg by subcutaneous injection on days 1, 3, 5 & 7
  Interventions: Drug: Interferon-Beta
- Aspirin (ASA) (Experimental): Outpatients:
  75 to 100 mg once daily for 28 days.
  Inpatients:
  75 to 100 mg once daily for 28 days
  Interventions: Drug: Aspirin
- Rivaroxaban (Experimental): Inpatients Only:
  2.5 mg twice daily for 28 days.
  Interventions: Drug: Rivaroxaban
- Usual Care (Control) (No Intervention): Outpatients and Inpatients: No constraints for treating physicians on the therapies within the standard of care arm. All key co-interventions will be documented.

INTERVENTIONS:
Drug: Colchicine — oral medication
  Arms: Colchicine
Drug: Interferon-Beta — subcutaneous injection
  Arms: Interferon Beta [This arm is now closed to recruitment]
Drug: Aspirin — oral medication
  Arms: Aspirin (ASA)
Drug: Rivaroxaban — oral medication
  Arms: Rivaroxaban

SUMMARY:
ACT is a randomized clinical trial to assess therapies to reduce the clinical progression of COVID-19.

DETAILED DESCRIPTION:
The ACT COVID-19 program consists of two parallel trials testing the effects of interventions in complementary populations in outpatients and inpatients.

In the outpatient study, symptomatic patients in the community who are COVID-19 positive and at high risk of disease progression: colchicine compared with control (anti-inflammatory); and ASA compared with control (anti-thrombotic); using a 2 x 2 factorial design. The primary outcome for colchicine vs. control is the composite of hospitalization or death. The primary outcome for ASA vs. control is the composite of hospitalization, death, or major thrombosis [myocardial infarction(MI), stroke, acute limb ischemia(ALI), or pulmonary embolism (PE)].

For inpatients, in symptomatic patients who are COVID-19 positive and who are hospitalized: colchicine is compared with control (anti-inflammatory), and the combination of ASA and rivaroxaban is compared with control (anti-thrombotic); using a 2 x 2 factorial design. The primary outcome for colchicine vs. control is the composite of high flow oxygen, mechanical ventilation, or death. The primary outcome for the combination of ASA and rivaroxaban vs. control is the composite of high flow oxygen, mechanical ventilation, death, or major thrombosis (MI, stroke, ALI, or PI).

*The Inpatient study previously also included a comparison of Interferon-β with control in a 2x2x2 design. The Interferon-β arm was closed to recruitment in November 2020.

ELIGIBILITY:
Outpatient trial:

Inclusion criteria:

1. Symptomatic and laboratory-confirmed diagnosis of COVID-19.
2. Age ≥ 30 years.
3. High risk: either age ≥70 or one of the following: male; obesity (BMI ≥30); chronic cardiovascular, respiratory or renal disease; active cancer; diabetes.
4. Within 7 days (ideally 72 hours) of diagnosis, or worsening clinically.

Exclusion criteria:

1. General: advanced kidney disease; advanced liver disease; pregnancy (known or potential) or lactation.
2. Colchicine: allergy or planned use; current or planned use of cyclosporine, verapamil, HIV protease inhibitor, azole antifungal, or macrolide antibiotic (except azithromycin).
3. ASA: allergy; high risk of bleeding, current or planned use of other anti-thrombotic drugs (e.g., P2Y12 inhibitors, direct oral anticoagulants, vitamin K antagonists, heparins)

Inpatient trial:

Inclusion criteria:

1. Symptomatic and laboratory-confirmed diagnosis of COVID-19.
2. Age ≥18 years.
3. Within 72 hours (ideally 24 hours) of admission, or worsening clinically.

Exclusion criteria:

1. General: advanced kidney disease; advanced liver disease, pregnancy (known or potential) or lactation, already ventilated for >72 hours.
2. Colchicine: allergy or planned use; current or planned use of cyclosporine, verapamil, HIV protease inhibitors, azole antifungals, or macrolide antibiotics (except azithromycin).
3. ASA and rivaroxaban: allergy; high risk of bleeding; estimated GFR <15 ml/min; current or planned use of P2Y12 inhibitors or therapeutic doses of anticoagulants* (e.g., direct oral anticoagulants, vitamin K antagonists, heparin, LMWH), current or planned use of strong inhibitors of both CYP 3A4 and P-gp (e.g., lopinavir/ritonavir, carbamazepine, ketoconazole). *Note that prophylactic doses of anticoagulants can be used in patients who are randomized to control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6667 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Outpatient trial - Colchicine vs. control: Time from randomization to first occurrence of the composite of hospitalization or death | 45 days post randomization
Outpatient trial - Aspirin vs. control: Time from randomization to first occurrence of the composite of hospitalization, death or major thrombosis (MI, stroke, ALI, or PE) | 45 days post randomization
Inpatient trial - Colchicine vs. control: Time from randomization to first occurrence of the composite of high flow oxygen, mechanical ventilation, or death | 45 days post randomization
Inpatient trial - Aspirin and Rivaroxaban vs. control: Time from randomization to first occurrence of the composite of high flow oxygen, mechanical ventilation, death or major thrombosis (MI, stroke, ALI, or PE) | 45 days post randomization

SECONDARY OUTCOMES:
Outpatient trial - Aspirin vs. control: Time from randomization to first occurrence of any thrombosis (MI, stroke, ALI, PE, or DVT) | 45 days post randomization
Inpatient trial - Colchicine vs. control: Time from randomization to first occurrence of the composite of high flow oxygen, mechanical ventilation, or respiratory death | 45 days post randomization
Inpatient trial - Aspirin vs. control: Time from randomization to first occurrence of the composite of high flow oxygen, mechanical ventilation, or respiratory death | 45 days post randomization
Inpatient trial - Aspirin vs. control: Time from randomization to first occurrence of any thrombosis (MI, stroke, ALI, PE, or DVT) | 45 days post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, MD PhD, Principal Investigator — Population Health Research Institute; Emilie Belley-Cote, MD PhD, Principal Investigator — Population Health Research Institute; John Eikelboom, MBBS MSc, Principal Investigator — Population Health Research Institute
Locations (66):
- Brazil (10):
  - Hospital Adventista de Manaus, Manaus, Amazonas
  - Hospital das Clinicas de Vitoria (Hospital Universitario Cassiano Antonio Moraes), Vitória, Espírito Santo
  - Prodal Saude S/A, Salvador, Estado de Bahia
  - Ubermed Serviços em Saúde Eireli - Hospital São Domingos, Uberaba, Minas Gerais
  - Hospital de Clínicas da Universidade Federal de Uberlândia, Uberlândia, Minas Gerais
  - Hospital Universitario Julio Muller, Cuiabá, Mount
  - Instituto Tacchini de Pesquisa em Saude / Hospital Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Hospital Universitario Prof. Dr. Horacio Carlos Panepucci da Universidade Federal de Sao Carlos (HU-UFSCar), São Carlos, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Santa Casa de Votuporanga, Votuporanga, São Paulo
- Canada (11):
  - CardiAI Inc., Calgary, Alberta
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Halton Healthcare/Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - Niagara Health System-St. Catharine's, St. Catharines, Ontario
  - Toronto Western Hospital Family Health Team, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - Woodstock Hospital, Woodstock, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - CIUSSS de L'est-de-l'ile de Montreal, Hopital Maisonneuve-Rosemont, Montreal, Quebec
- Colombia (3):
  - Biomelab SAS, Barranquilla, Atlántico
  - Clinica de la Costa LTDA, Barranquilla, Atlántico
  - Instituto de Neumologico del Oriente, Bucaramanga, Santander Department
- Ecuador (5):
  - Unicormed, Guayaquil, Guayas
  - Hospital de Especialidades Eugenio Espejo, Quito, Pichincha
  - Hospital Enrique Garces, Quito, Pichincha
  - Hospital General Pablo Arturo Suarez, Quito, Pichincha
  - Oncoambato, Ambato, Tungurahua Province
- Egypt (5):
  - Giza Chest Hospital, Giza, Cairo Governorate
  - Fayoum University Hospital, Al Fayyum
  - Abbasia Chest Hospital, Cairo
  - Abbasia Fever Hospital, Cairo
  - National Hepatology and Tropical Medicine Research Institute, Cairo
- India (7):
  - St. John's Medical College and Hospital, Bangalore, Karnataka
  - Bharathi Hospital and Research Center, Pune, Maharashtra
  - Sanjeevan Hospital, Pune, Maharashtra
  - Sidhu Hospital Pvt.Ltd, Dorāha, Punjab
  - SRM Medical College Hospital & Research Center, Chengalpattu, Tamil Nadu
  - AIG Hospital, Hyderabad, Telangana
  - KIMS, Secunderabad, Telangana
- Nepal (6):
  - Chitwan Medical College, Bharatpur-10, Bagmati
  - Sahid Gangalal National Heart Center, Kathmandu, Bagmati
  - Province Hospital, Karnali Province, Surkhet, Karnali
  - Mechi Zonal Hospital, Bhadrapur, Province No. 1
  - Koshi Zonal Hospital, Biratnagar, Province No. 1
  - B.P. Koirala Institute of Health Sciences, Kathmandu, Province No.1
- Pakistan (3):
  - Aga Khan University Hospital, Karachi, Sindh
  - Jinnah Postgraduate Medical Center, Karachi, Sindh
  - Tabba Heart Institute, Karachi, Sindh
- Philippine General Hospital, Manila, National Capital Region, Philippines
- Russia (9):
  - Central City Clinical Hospital No. 24, Yekaterinburg, Sverdlovsk Oblast
  - State Budgetary Health Care Institution of Sverdlovsk region "Central city clinical hospital # 6 Ekaterinburg", Yekaterinburg, Sverdlovsk Oblast
  - Tver State Medical University, Tver', Tver Oblast
  - Voronezh State Medical University named after N.N. Burdenko, Voronezh, Voronezh Oblast
  - Altai Regional Center for Medical Prevention, Barnaul
  - City Clinical Hospital No. 15 named after O.M. Filatova, Moscow
  - National Medical Research Center for Therapy and Preventive Medicine, Moscow
  - City Clinical Hospital No. 3, Nizhny Novgorod
  - Rostov State Medical University, Rostov-on-Don
- South Africa (3):
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - University of Cape Town- Groote Schuur Hospital, Cape Town, Western Cape
  - TASK Eden, George, Western Cape
- United Arab Emirates (3):
  - Hatta Hospital, Hatta, Dubai
  - Rashid Hospital, Dubai Health Authority, Dubai
  - Thumbay Hospital Dubai, Dubai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818
- [Derived] Eikelboom JW, Jolly SS, Belley-Cote EP, Whitlock RP, Rangarajan S, Xu L, Heenan L, Bangdiwala SI, Luz Diaz M, Diaz R, Yusufali A, Kumar Sharma S, Tarhuni WM, Hassany M, Avezum A, Harper W, Wasserman S, Almas A, Drapkina O, Felix C, Lopes RD, Berwanger O, Lopez-Jaramillo P, Anand SS, Bosch J, Choudhri S, Farkouh ME, Loeb M, Yusuf S. Colchicine and the combination of rivaroxaban and aspirin in patients hospitalised with COVID-19 (ACT): an open-label, factorial, randomised, controlled trial. Lancet Respir Med. 2022 Dec;10(12):1169-1177. doi: 10.1016/S2213-2600(22)00298-3. Epub 2022 Oct 10. PMID 36228641
- [Derived] Eikelboom JW, Jolly SS, Belley-Cote EP, Whitlock RP, Rangarajan S, Xu L, Heenan L, Bangdiwala SI, Tarhuni WM, Hassany M, Kontsevaya A, Harper W, Sharma SK, Lopez-Jaramillo P, Dans AL, Palileo-Villanueva LM, Avezum A, Pais P, Xavier D, Felix C, Yusufali A, Lopes RD, Berwanger O, Ali Z, Wasserman S, Anand SS, Bosch J, Choudhri S, Farkouh ME, Loeb M, Yusuf S. Colchicine and aspirin in community patients with COVID-19 (ACT): an open-label, factorial, randomised, controlled trial. Lancet Respir Med. 2022 Dec;10(12):1160-1168. doi: 10.1016/S2213-2600(22)00299-5. Epub 2022 Oct 10. PMID 36228639
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014